CLINICAL TRIAL: NCT03872804
Title: Punch Minigraft Versus Transverse Needling or Combination of Both in Treatment of Non-Segmental Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Omneya abd el aziz abd el rehim el zagh, Principle investigator, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlexandriadermaU
Record Dates: First submitted 2019-03-06; First posted 2019-03-13 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Vitiligo
Keywords: Vitiligo; Punch graft; Oral pulse steroid; Transverse needling
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitiligo patient (Experimental): Patient has at least 4 patches , one of them will be treated by autologous punch graft , second one by transverse needling , third one with minigraft followed by needling , fourth one as control under treatment with oral pulse steroid with narrow band .
  Interventions: Procedure: Autologous punch mini grafts:; Procedure: Transverse needling; Procedure: Punch minigrafts followed by transverse needling; Other: Oral pulse steroid with narrow band

INTERVENTIONS:
Procedure: Autologous punch mini grafts: — Under local anesthesia, multiple 1mm holes will be made in the depigmented treatment area using 1mm punch graft instrument inserted to a depth of 2-4 mm to remove a small column of depigmented skin that is to be discarded. The punches will be situated at or very close to the border of the lesion to avoid leaving an achromic fissure and will be separated by 5-8 mm distance from each other.
  On the donor area mostly is the gluteal area, punches will be harvested using the same sized punches very close to each other so that maximum number of grafts can be taken from a small area.
  Then the harvested-punch minigrafts will be inserted into the recipient chambers, pressed firmly by saline soaked gauge for hemostasis and secured by sterile strips or a compression bandage if applicable.
Procedure: Transverse needling — Needling will be done for selected treatment patch using a 30 G disposable insulin syringe, going from the pigmented margins of the lesion into the vitiliginous patch, Position of the needle will be kept close to the dermoepidermal junction and movement will be from normal skin towards the lesion. Needle pricks may lead to oozing of a small drop of blood which will be managed by physical pressure. No dressings will be needed. The procedure will be repeated for selected lesions weekly for a duration of 3 months.
Procedure: Punch minigrafts followed by transverse needling — In a third lesion, punch minigrafts will be done as mentioned in line 1 and will be left to stabilize for 3 months then transverse needling will be done weekly for the margins of the lesion as well as the areas of the punch grafts toward the vitiliginous area.
Other: Oral pulse steroid with narrow band — * A fourth lesion will be chosen as a control lesion, to which no surgical treatment will ba attempted.
  * All lesions will receive NB-UVB therapy according to standard protocol twice weekly and the patients will continue on the oral mini pulse dexamethasone at 2.5 mg dose for two consecutive days weekly all through the study period

SUMMARY:
This study is to evaluate the effectiveness and tolerability of autologous punch minigraft, transverse needling technique or combination of both followed by narrow band ultraviolet B phototherapy (311 nm) in the treatment of patients with stable non-segmental vitiligo lesions.

DETAILED DESCRIPTION:
Vitiligo is a common pigmentary cutaneous disorder occurring with an incidence of 1-2% worldwide, without predilection for sex or race.

The disease is characterized by gradual loss of the normal color of the skin resulting from melanin pigment loss due to the underlying destruction of the melanocyte.

Vitiligo is a multifactorial disorder with many theories explaining its pathogenesis such as autoimmunity, self-destructing mechanisms,neural mediators, biochemicals,an imbalance of epidermal cytokines and genetic factors.

Vitiligo is not a life-threatening disease,but it may cause a major social and emotional distress with significant impairment in the quality of life.

Clinically; vitiligo is classified into segmental, non-segmental and unclassified vitiligo .Non-segmental includes generalized, acrofacial,universal, mucosal (more than one mucosal site) , mixed (associated with segmental vitiligo) and other rare variants. Segmental vitiligo includes uni- ,bi- or pluri-segmental subtypes. Unclassified includes focal or mucosal (one site) subtypes.

Treatment options for vitiligo include attempting repigmentation of affected areas,

depigmentation of non-involving skin or camouflage if neither is effective.Repigmentation could be attempted using medical therapy, surgical modalities.

Topical medications include corticosteroids or calcineurin inhibitors.Ultraviolet radiation therapy, such as narrow-band ultraviolet B light (NB-UVB), is also widely used. It is minimally invasive, has few adverse effects and provides a good response rate. Excimer laser or light has become available for use recently, and favorable treatment results have been reported.

When medical treatments are ineffective, surgical treatment is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>16 years old) of either gender having stable non segmental vitiligo, that is resistant to other lines of repigmentation therapy.
* Lack of progression of old lesions with the past 6 months.
* No development of new lesions
* Absence of history of koebner phenomenon.
* Absence of confetti lesions or hypopigmented lesions within the past 6 months.
* Presence of repigmentation of depigmented areas by medications or spontaneously in the past 6 months.
* While resistance to therapy will be judged after receiving standard protocol of NB-UVB together with oral mini pulse dexamethasone at a dose of 2.5 mg on two consecutive weekly days for 3 months.
* Patients having lesions showing absence or poor repigmentation after this regiment will be considered resistant to medical repigmentation and indicated to surgery.

Exclusion Criteria:

* Cases of active, progressive disease lacking criteria of stability previously mentioned.
* Patients with segmental or universal vitiligo covering more than 70% body surface area.
* Patients with known associated autoimmune diseases, bleeding tendency, current or history of skin neoplasia, photosensitive disorders or any contraindications to corticosteroids therapy.
* Patients with tendency towards hypertrophic scars or keloid formation.
* Pregnant female and lactating mothers.
* Patients with emotional and psychological instability.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of repigmentation | 6 months
  Assessments of repigmentation will be performed by two blinded dermatologists using a 5-point scale; grade 0 (no repigmentation), grade 1 (1%-5%), grade 2 (6%-25%), grade 3 (26%-50%), grade 4 (51%-75%) and grade 5 (76%-100%)
Evaluation of Type, pattern and extent of repigmentation. | 6 months
  Serial photography will be done to evaluate type, pattern and extent of repigmentation.
Digital assessment of the size of the lesion and of the depigmented versus repigmented area | 6 months
  Digital assessment of the size of the lesion and of the depigmented versus repigmented area using Adobe photoshop software

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Ibrahiem farid amin, Ph.D, Study Director — Assistant Professor of dermatolog Faculty of Medicine. University of Alexandria.; Magdy Abd el aziz ragab, Ph.D, Study Director — Professor of Dermatlolgy, Faculty of Medicine. University of Alexandria.
Locations (1):
- Omneya abd el aziz el zagh, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT03872804/Prot_000.pdf